CLINICAL TRIAL: NCT06689488
Title: Assessment of the Safety and Performance of the AB1 Electrosurgical System for Bronchoscopic Microwave Ablation of Lung Tissue in Surgical Candidates
Brief Title: Bronchoscopic Microwave Ablation of Lung Tissue in Surgical Candidates
Acronym: AB1MALTISC
Status: Recruiting | Type: Observational
Sponsor: Creo Medical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-GTD-AB1-003
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: Bronchoscopy; Ablation; Microwave; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Resected lung tissue and blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Microwave ablation: Patients with a malignant lung nodule who are candidates for surgical resection.
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Bronchoscopy and microwave ablation prior to surgical resection.

SUMMARY:
The overall purpose of this study is to characterise the clinical safety and performance of the Creo Medical MicroBlate™ Flex AB1 instrument in patients with pathologically confirmed malignancy eligible for surgical resection of their nodule, receiving bronchoscopic ablation prior to surgery.

DETAILED DESCRIPTION:
This is a post-market, prospective, single-arm, multicentre, open-label, non-randomised study which will enrol up to 30 subjects in total (plus replacements if required due to drop out).

Prospective patients must have a histopathological-confirmed malignant lung lesion and be candidates for surgical resection. After being informed about the study and potential risks, all patients giving their written informed consent will undergo a screening visit to determine eligibility for study entry.

The study consists of two (2) stages (Stage A and Stage B). Stage A consists of the ablation and surgical resection being performed concurrently on Day 0 within a single procedure. Stage B consists of the ablation and the surgical resection being performed in separate procedures. The surgical resection will occur between Day 7 and Day 21, post-ablation, inclusive of those days. The aim is to follow local guidelines for treatment of lung cancer.

Patients undergoing Stage A will be released from the study at point of standard of care discharge from hospital post-surgery and will not be followed as part of the study (patients will receive SoC follow-up and care post release from study).

Patients undergoing Stage B will have evaluations at follow-up visits conducted at 7 (+/-3) days (via phone call) post ablation and prior to the surgical resection procedure. Stage B patients will be released from the study at point of standard of care discharge from hospital post-surgery and will not be followed as part of the study (patients will receive SoC follow-up and care post release from study).

ELIGIBILITY:
Inclusion Criteria:

Patients who:

1. Have signed informed consent.
2. Subject is willing and able to comply with all aspects of the treatment and evaluation schedule.
3. Are ≥ 18 years old.
4. Have lung lesion(s)/nodule(s) which are histopathological-confirmed as cancer.
5. Have soft tissue lung lesion(s):

   * ≤ 30 mm in the largest dimension of the pulmonary window for Stage A.
   * ≤ 20 mm in the largest dimension of the pulmonary window for Stage B.
6. Are candidates for surgical resection as determined by a multi-disciplinary team (MDT) or tumour board.
7. Greater than 10 mm of tumour-free lung parenchyma between target tumour and pleura or fissure.
8. Subject is willing and able to comply with the study protocol requirements.
9. Are assigned an ASA (American Society of Anaesthesiologists) score of ≤ 3 or the patient is deemed fit for general anaesthesia.

Exclusion Criteria:

Patients who:

1. Have target nodule(s) within the International Association for the Study of Lung Cancer (IASLC) "Central Zone" (including bronchial tree, major vessels, heart, oesophagus, spinal cord, and phrenic & laryngeal nerves).
2. Are pregnant or breast feeding, as determined by standard site practices.
3. Have participated in an investigational drug or device research study within 30 days of enrolment that would interfere with this study.
4. Have a physical or psychological condition that would impair study participation or jeopardise the safety or welfare of the subject.
5. Have an expected survival less than 12 months.
6. Have bleeding diathesis, uncorrectable coagulopathy, or platelet count ≤ 100 x 10^9/L.
7. Have an implantable device, including pacemakers or other electronic implants.
8. Have known pulmonary hypertension (PASP [pulmonary artery systolic pressure] >50mmHg).
9. Who are currently prescribed anticoagulants, clopidogrel or other platelet aggregation inhibitors which can´t be stopped or temporarily withheld.
10. Subject had a prior pneumonectomy.
11. Diagnosis of Small Cell Lung Cancer.
12. Any patient with clinically significant interstitial lung disease in the zone of planned ablation.
13. Subject had a therapeutic intervention (e.g., SBRT) within same lobe as the target lesion.
14. Subjects currently undergoing or underwent chemotherapy, systemic immunosuppressive treatment, or radiotherapy within 3 months of planned Study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population going through lung cancer screening at investigative sites.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Day 0, day of ablation procedure up to initiation of surgical resection procedure.
  Stage A - Ablate (Day 0) & Resect (Day 0) Identification of serious device-related intra-procedural adverse events related to the use of the AB1 system on Day 0 prior to surgical resection defined by the initial skin incision (number and nature of serious adverse events, both device and procedure related, will be identified).
Primary Safety Endpoint | Day 7-21, post ablation procedure up to initiation of surgical resection procedure.
  Stage B - Ablate (Day 0) & Resect (Resection Day 7-21) Identification of serious device-related adverse events related to the use of the AB1 system from day 0 up to initiation of surgical resection procedure (number and nature of serious adverse events, both device and procedure related, will be identified).
Primary Performance (Efficacy) Endpoint | Up to 1 week post ablation procedure.
  Initial technical success, defined as successful bronchoscopic access by the AB1 instrument of the target tissue, delivery of scheduled microwave energy to the target tissue (per pre-specified target) and confirmed ablation as evidenced by macroscopic assessment post-surgical resection of the ablated lesion.

SECONDARY OUTCOMES:
Secondary Performance (Efficacy) Endpoints - Assessment/visualization/quantification of the dimensions of the ablated tissue including assessment of margin relative to lesion | Up to 1 week post ablation procedure.
  Dimensions of the ablated tissue to confirm, correct or add to the IFU-reported relationship between AB1 ablation time and dimensions and volume of the ablated tissue, per pre-specified target.
Secondary Performance (Efficacy) Endpoints - Assessment/visualization/quantification of the dimensions of the ablation observed within the post-ablation CT | Up to 1 week post ablation procedure.
  Dimensions of the ablated tissue as evidenced on the post ablation CT.
Secondary Performance (Efficacy) Endpoints - Procedural Time | Up to 1 week post ablation procedure.
  Procedural time to be captured in the electronic case report form (eCRF).
Secondary Performance (Efficacy) Endpoints - Assessment of ease of system use (clinician questionnaires) | Up to 1 week post ablation procedure.
  Questionnaires to be completed by clinicians, rating their responses on a Likert scale of 1 to 7, with 1 being "extremely clear/easy" and 7 being "extremely difficult".

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD, Principal Investigator — Amsterdam University Medical Centres
Locations (1):
- Amsterdam University Medical Centres, Location AMC, Meibergdreef 9, Amsterdam, The Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Summary aggregate information will be published in a PRJA at the conclusion of the study.

REFERENCES:
- [Background] Covey AM, Gandhi R, Brody LA, Getrajdman G, Thaler HT, Brown KT. Factors associated with pneumothorax and pneumothorax requiring treatment after percutaneous lung biopsy in 443 consecutive patients. J Vasc Interv Radiol. 2004 May;15(5):479-83. doi: 10.1097/01.rvi.0000124951.24134.50. PMID 15126658
- [Background] Licker MJ, Widikker I, Robert J, Frey JG, Spiliopoulos A, Ellenberger C, Schweizer A, Tschopp JM. Operative mortality and respiratory complications after lung resection for cancer: impact of chronic obstructive pulmonary disease and time trends. Ann Thorac Surg. 2006 May;81(5):1830-7. doi: 10.1016/j.athoracsur.2005.11.048. PMID 16631680
- [Background] Boffa DJ, Allen MS, Grab JD, Gaissert HA, Harpole DH, Wright CD. Data from The Society of Thoracic Surgeons General Thoracic Surgery database: the surgical management of primary lung tumors. J Thorac Cardiovasc Surg. 2008 Feb;135(2):247-54. doi: 10.1016/j.jtcvs.2007.07.060. Epub 2007 Dec 21. PMID 18242243
- [Background] Chen H, Senan S, Nossent EJ, Boldt RG, Warner A, Palma DA, Louie AV. Treatment-Related Toxicity in Patients With Early-Stage Non-Small Cell Lung Cancer and Coexisting Interstitial Lung Disease: A Systematic Review. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):622-631. doi: 10.1016/j.ijrobp.2017.03.010. Epub 2017 Mar 15. PMID 28581404
- [Background] SABR UK Consortium. "Stereotactic Ablative Body Radiation Therapy (SABR): A Resource." Version 6.1. January 2019
- [Background] Chang et al The Lancet Oncology 2015 Vol 16, Issue 6, 630 - 637